CLINICAL TRIAL: NCT00043875
Title: A Double-Blind, Placebo-Controlled, Add-On Clinical Trial of the Safety, Pharmacokinetics and Efficacy of Lamictal in Pediatric Age Subjects (1-24 Months)
Brief Title: Pediatric Epilepsy Trial in Subjects 1-24 Months
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LAM20006
Record Dates: First submitted 2002-08-14; First posted 2002-08-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Epilepsy
Keywords: partial seizures; pediatric; epilepsy
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: lamotrigine

SUMMARY:
This study is being conducted to evaluate the effectiveness and safety of LAMICTAL added to the current therapy of pediatric patients age 1-24 months old with partial seizures. The medication used in this study has been approved by FDA for the adjunctive treatment of partial seizures in patients 2 years and older.

ELIGIBILITY:
INCLUSION CRITERIA:

* Have a confident diagnosis of epilepsy
* Must be experiencing 4 or more reliably detectable partial seizures per month while receiving at least 1 anti-epileptic drug (AED)
* Must weigh at least 7 lbs if currently receiving enzyme inducing antiepileptic drugs (EIADs) OR weigh at least 15 lbs if currently receiving non-enzyme inducing antiepileptic drugs (non-EIADs)
* Have no underlying chronic metabolism problems
* Have normal lab results
* Have a normal electrocardiogram (ECG)

EXCLUSION CRITERIA:

* Have a diagnosis of severe, progressive myoclonus.
* Have seizures not related to epilepsy.
* Have previously demonstrated sensitivity or allergic reaction to the study drug or its related compounds.
* Have progressive or unstable condition of the nervous system.
* Used experimental medication within 30 of enrollment into the study.
* Have any significant, chronic heart, kidney, liver or stomach/intestinal (GI) condition.
* Current use of the medication felbamate.
* Current use of adrenocorticotrophic hormone (ACTH).
* Following a ketogenic diet.
* Receiving vagal nerve stimulation (VNS).

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 177 (Actual)
Dates: Start 2000-05; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
The efficacy of LAMICTAL add-on therapy will be measured by the proportion of subjects who meet escape criteria during the Double-Blind Phase. | 36 Months

SECONDARY OUTCOMES:
Time to escape patterns in Double-Blind phase. Reduction in partial seizure frequency at end of Open-Label Phase. Investigators' global evaluation of subjects' status at end of Open-Label and Double-Blind Phases; Standard pharmacokinetics; Adverse Events | 36 Months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (63):
- United States (32):
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Stanford, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Saint Paul, Minnesota
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Cherry Hill, New Jersey
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
- Australia (4):
  - GSK Investigational Site, South Brisbane, Queensland
  - GSK Investigational Site, Parkville, Melbourne, Victoria
  - GSK Investigational Site, West Heidleberg, Melbourne, Victoria
  - GSK Investigational Site, Perth, Western Australia
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- GSK Investigational Site, Reims, France
- Hungary (4):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Miskolc
  - GSK Investigational Site, Szeged
- Italy (6):
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Mantova, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Messina, Sicily
  - GSK Investigational Site, Padua, Veneto
- GSK Investigational Site, Riga, Latvia
- GSK Investigational Site, Beirut, Lebanon
- GSK Investigational Site, Kaunas, Lithuania
- Netherlands (3):
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Utrecht
- Portugal (3):
  - GSK Investigational Site, Coimbra
  - GSK Investigational Site, Lisbon
  - GSK Investigational Site, Porto
- Slovakia (3):
  - GSK Investigational Site, Banská Bystrica
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Prešov
- GSK Investigational Site, Las Palmas de Gran Canaria, Spain
- GSK Investigational Site, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: LAM20006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: LAM20006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: LAM20006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: LAM20006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: LAM20006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: LAM20006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: LAM20006 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register